CLINICAL TRIAL: NCT01356342
Title: Immunogenicity and Safety of a Trivalent Inactivated Influenza Vaccine, Formulation 2010-2011, in Healthy Subjects Aged Over 6 Months Old to 18 Years Old
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Adimmune Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FLU10T11B
Record Dates: First submitted 2011-05-16; First posted 2011-05-19 (Estimated); Last update posted 2012-12-28 (Estimated); Status verified 2012-12

CONDITIONS: Influenza
Keywords: Influenza; Vaccine; Immunogenicity
MeSH Terms: conditions — Influenza, Human

ARMS (3):
- AdimFlu-S 2010-2011, 6 months~<3 years (Experimental)
  Interventions: Biological: AdimFlu-S 2010-2011, inactivated
- AdimFlu-S 2010-2011,3~<9 years (Experimental)
  Interventions: Biological: AdimFlu-S 2010-2011, inactivated
- AdimFlu-S 2010-2011,9~<18 years (Experimental)
  Interventions: Biological: AdimFlu-S 2010-2011, inactivated

INTERVENTIONS:
Biological: AdimFlu-S 2010-2011, inactivated — The vaccine contains not less than 90 μg haemagglutinin (HA) per mL. Per mL contains the following three strains: A/California/7/2009 (H1N1)30 μg/mL;A/Perth/16/2009 (H3N2)30 μg/mL;B/Brisbane/60/2008 30 μg/mL
  6 months~<3 years;0.25 mL per injection2 injections at 4 weeks apart
  3~<9 years;0.5 mL per injection2 injections at 4 weeks apart
  9~<18 years;0.5 mL per injection1 injections

SUMMARY:
This is an open study of the use of AdimFlu-S (2010-2011 season) vaccine in young subjects aged between 6 months old to 18 years old. All participants will be divided into three age cohorts. First, participants aged 6 through < 36 months will receive 2 doses of 0.25 mL vaccine separated by 4 weeks. Second, participants aged 3 through < 9 years will receive 2 doses of 0.5 mL vaccine separated by 4 weeks. Third, participants aged 9 through < 18 years will receive one dose of 0.5 mL vaccine. Safety outcomes included immediate reactions at the time of vaccination, solicited local and systemic reactions within 7 days after each vaccination, unsolicited adverse events, and serious adverse events. Sera prepared from blood samples will be collected from each subject immediately prior to, and 4 weeks after each vaccination. Anti-hemaglutinin (HA) antibody titers will be determined using the WHO haemaglutination inhibition reference technique. The analysis will be observer-blinded. All participants will be followed, either by clinical visit or by telephone contact, for 6 months after the first vaccination for safety reasons.

ELIGIBILITY:
Inclusion Criteria:

* Boys or girls and aged 6 months old to 18 years old on the day of first vaccination;
* Subject and/or parents(s)/legal guardian(s) must be willing to comply with planned study procedures and be available for all study visits;
* Subject must be in good physical health on the basis of medical history, physical examination;
* Subject and/or parents(s)/legal guardian(s) must read and signed the study-specific informed consent prior to initiation of any study procedure.

Exclusion Criteria:

* Subjects received influenza vaccine (Trivalent and/or A(H1N1)) within the previous 6 months;
* History of hypersensitivity to eggs or egg protein or similar pharmacological effects to study medication;
* Personal or family history of Guillain-Barré Syndrome;
* An acute febrile illness within 1 week prior to vaccination;
* Current upper respiratory illness (URI), including the common cold or nasal congestion within 72 hours;
* Subjects with influenza-like illness as defined by the presence of fever (temperature ³38ºC) and at least two of the following four symptoms: headache, muscle/joint aches and pains (e.g. myalgia/arthralgia), sore throat and cough;
* Female subjects who are pregnant, lactating or likely to become pregnant during the study; Women of childbearing potential disagree to use an acceptable method of contraception (e.g., hormonal contraceptives, IUD, barrier device or abstinence) throughout the study;
* Treatment with an investigational drug or device, or participation in a clinical study, within 3 months before consent;
* Immunodeficiency, immunosuppressive or household contact with immunosuppression;
* History of wheezing or bronchodilator use within 3 months prior to study vaccine;
* Receipt of live virus vaccine within 1 month prior to study vaccine or expected receipt vaccination before the last blood sampling for immunogenicity evaluation;
* Receipt of any inactivated vaccine within 2 weeks prior to study vaccination or expected receipt vaccination before the last blood sampling for immunogenicity evaluation;
* Receipt of any blood products, including immunoglobulin in the prior 3 months;
* Underlying condition in the investigators' opinion may interfere with evaluation of the vaccine;
* Significant chronic illness for which inactivated influenza vaccine is recommended or commonly used.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 181 (Actual)
Dates: Start 2010-07; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
The primary objective is to evaluate the immunogenicity profiles for influenza virus vaccine strains (2010-2011 season) of the AdimFlu-S manufactured by Adimmune Corporation. | Serum samples will be obtained prior to vaccination (baseline), and 4 weeks after each vaccination.
  Serum samples will be obtained prior to vaccination, and 4 weeks after each vaccination. Serum samples will be tested for anti-hemaglutinin (HA) antibodies by hemagglutinaton inhibition (HAI), and assays will be performed at Adimmune Corporation designated central laboratory. Subjects will be considered to be seronegative if serum HAI titer<1:10. The seroconversion is defined as the post-vaccination serum at least 40 for whom had negative pre-vaccination or a fourfold or greater increase in HAI titers in subjects who had positive pre-vaccination serum.

SECONDARY OUTCOMES:
The secondary objective is to evaluate the safety and tolerability profiles including the presence or absence of the pre-specified reactogenicity events and other serious/non-serious adverse events of the AdimFlu-S manufactured by Adimmune Corporation. | Safety data will consist of reactogenicity, serious and non-serious adverse events throughout the study, including 7 days after each dose of study vaccine. Vital signs and physical examination will be performed at each clinic visit.
  Reactogenicity events are pre-specified adverse events systematically recorded on diary cards (a grid of check boxes for each event and each day) during the immediate post-vaccination period by all participants. In general, reactogenicity events will be recorded for 7 days after each vaccination. The selection of the events to be collected systematically is based on events expected to occur with wild-type influenza infection.